CLINICAL TRIAL: NCT04723511
Title: Effect of Global Postural Reeducation on Functional Abilities, Stability of Sense of Position, Cognitive Abilities and Treatment Satisfaction in Patients With Forward Head Posture
Brief Title: Effects of Global Postural Reeducation on Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Abu-Taleb, Principal investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002671
Record Dates: First submitted 2021-01-15; First posted 2021-01-25 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Forward Head Posture
Keywords: Forward Head Posture; Global Postural Re-education; Kendall Exercises; Rounded Shoulders; Postural Correction; Myofascial chains

STUDY DESIGN:
Who Masked: Participant
Masking Description: The enrolled participants will be masked (single blind study) and randomly assigned into two groups without being informed whether they are in the control or the study(experimental) group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPR (Experimental): participants in this group receive global postural reeducation technique+ Kendall exercises
  Interventions: Other: Global Postural Re-education; Other: Kendall exercises
- Kendall (Active Comparator): Kendall exercises
  Interventions: Other: Kendall exercises

INTERVENTIONS:
Other: Global Postural Re-education — treatment techniques include corrective exercises both local and global to correct forward head posture.
  first session will be to educate participants on the treatment sequence. This will be a session of Kendall's exercises as described below. This will followed be by performing GPR techniques of Anterior Chain stretch in the supine frog-like position for 20 minutes followed by posterior chain stretch against the wall for another 20 minutes. This is repeated in the first 6 sessions. Starting from the seventh session the time of holding each position is decreased to 15 minutes and a third position (standing against the wall) is introduced and performed for 15 minutes. Starting from the eighth session fourth position of sitting on the floor position is introduced and performed for another 15 minutes. total of a session will then take about 90 minutes.
  Pre-treatment diaphragmatic release and deep breathing exercises are applied at the beginning of each session
  Arms: GPR
Other: Kendall exercises — exercises that correct upper crossed syndrome:
  The treatment sequence will be:
  a) Strengthen deep Cervical Flexors via Chin tucks. Repetition will be repeated 10 times for 5 sets.
  (b) Stretching the cervical extensors. This is held for 1 minute and repeated 5 times.
  (c) Strengthening shoulder retraction. Repetition will be repeated 10 times for 5 sets.
  (d) Stretching the pectoralis muscle. This is held for 1 minute and repeated 5 times.
  Exercises will be progressed as the sessions develop.

SUMMARY:
This study aims at investigating the effects of application of twelve sessions of Global Postural Re-education Technique (GPR) and Kendall Exercises (KE) on Craniovertebral angle (CVA), Gaze Angle (GA), Shoulders Angle (SA), Pain, functional abilities, Range of Motion, stability of sense of position, cervical muscle strength and endurance, Spinal mobility, and Chest Expansion.

DETAILED DESCRIPTION:
A sample of 43 participants with a CVA less than 50 degrees will be randomly assigned to one of the two groups either receiving global postural reeducation added to traditional Kendall exercises or a group that receives Kendall Exercises only. Treatment sessions will be continued for a total of 12 sessions with a rate of 3 sessions per week. The effect of these two treatments will be assessed by various variables including: forward head angle, Gaze Angle and Shoulder angle via photogrammetry and Kinovea App, Pain intensity (VAS), functional abilities via neck disability index (NDI), cervical Range of motion and sense of position stability by Cervical Range of Motion instrument (CROM), Spinal mobility and chest expansion by tape measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from forward head Posture (CVA less than 50 degrees)
* All subjects are medically stable and do not suffer from any other diseases which might affect the trial results.
* BMI (18-24)
* Patients willing and able to participate in this treatment program.
* At least a moderate user of English.

Exclusion Criteria:

* History of whiplash injury.
* Patients who have undergone spinal surgeries or spinal fixations.
* Patients with a neurologic deficit in their upper limbs, such as hypertonia, hypotonia, hyporeflexia, absence of reflex, and vertebral instability.

The patient underwent other physical therapy programs in the last three months.

- Excessive use of smart technology

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
craniovertebral angle | before and after 12 sessions
  the angle formed between a horizontal line and a line extending from ear meatus and C7

SECONDARY OUTCOMES:
Gaze Angle | before and after 12 sessions
  the angle formed between the line extending from the tragus of the ear to the canthus of the eye.
Shoulder Angle | before and after 12 sessions
  the angle formed between the line extending from C7 to acromion with horizontal line
Proprioceptive stability test | before and after 12 sessions
  By utilizing CROM testing the patients' sense of location precision
Spinal mobility | before and after 12 sessions
  Fingers to floor test using a tape measurement
Chest expansion | before and after 12 sessions
  Axillary and Xyphoid chest expansion by the tape measurement
Cervical muscle strength and endurance | before and after 12 sessions
  Biofeedback stabiliser is used to measure the maximum time the muscles could hold in addition to time the contraction of 50% maximum muscle contractionis maintained.
Neck disability index | before and after 12 sessions
  a scale that tests the effect of treatment on functional abilities of patients.
Pain intensity | before and after 12 sessions
  Visual analogue scale is given to participants to select their pain scale level.

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Abu-Taleb, MSc, Principal Investigator — Cairo University
Locations (1):
- Horus University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No
These data are case sensitive and considered confidential regarding my supervisors' opinion and participants' request , So, upon their request I prefer to not share individual participant data (IPD) with other researchers